CLINICAL TRIAL: NCT03670498
Title: A Double-blind, Parallel Cumulative Medical Device Pivotal Clinical Study to Assess the Safety and Efficacy of the 4 Channel NMES, Multi-center Prospective Study (Pilot Study)
Brief Title: The Safety and Efficacy of the 4 Channel NMES on Swallowing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1806/475-002
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Dysphagia
Keywords: stroke; cervical spinal cord injury
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 channel Electrical Stimulation(revised sequential) (Experimental): apply 4 channel electrical stimulation device with protocol Is a revised sequential activation protocol, it sequentially Rt. suprahyoid m (ch 1), Lt. suprahyoid m (ch 2), thyrohyoid m (ch 3), sternothyroid m (ch 4) with 4 channel electrical stimulation device.
  Interventions: Device: 4 channel Electrical Stimulation Device
- 2 channel Electrical Stimulation(classical) (Active Comparator): apply 2 channel electrical stimulation device with protocol Is a revised sequential activation protocol, it simultaneously suprahyoid m (ch 1), thyrohyoid m (ch 2) with 2 channel electrical stimulation device.
  Interventions: Device: 2 channel Electrical Stimulation Device

INTERVENTIONS:
Device: 4 channel Electrical Stimulation Device — electrical stimulation at muscles which related with deglutition
  Arms: 4 channel Electrical Stimulation(revised sequential)
Device: 2 channel Electrical Stimulation Device — electrical stimulation at muscles which related with deglutition
  Arms: 2 channel Electrical Stimulation(classical)

SUMMARY:
This study is a pilot study to prepare clinical trials to evaluate the safety and effectiveness of 4-channel electric stimulation therapy devices as a newly developed function for the treatment of dysphagia disorders.

The purpose of this study is to investigate the difference in 4ch NMES and 2ch NMES, And to obtain the values such as mean, standard deviation and so on, and to determine the number of subjects to be studied for clinical trials of validation permission in the future.

DETAILED DESCRIPTION:
* Design: Prospective study
* Inclusion criteria of patient group: who has a dysphagia symptom and confirmed by video-fluoroscopic swallowing study
* Intervention: Participants are divided into two group and applied electrical stimulation by a "Synchronized Electrical Stimulation Device(SESD)" in 4channel or 2channel Neuromuscular Electrical Stimulation.
* Main outcome measures: videofluoroscopic parameters, EQ-5D (EuroQoL-5D) questionnaire, II. M. D Anderson dysphagia inventory

ELIGIBILITY:
Inclusion Criteria:

* patient who do not belong to the criteria excluded for subjects aged 19 years or older
* Patient who is confirmed to be dysphagia by videofluoroscopy
* Patients who need clinical application of electrical stimulation therapy equipment for dysphagia. ex) stroke, cervical spinal cord injury
* Those voluntarily agreeing to the clinical trial

Exclusion Criteria:

* Patient who refuse inspection, do not agree
* Simple "Commend obey", first step is impossible
* When instructions can not be executed due to dementia, psychiatric disorders, etc.
* Dysphagia occurs due to respiratory failure, neck surgery, etc.,
* Pregnant women and lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-04 (Actual); Study Completion 2019-08-04 (Actual)

PRIMARY OUTCOMES:
videofluoroscopic dysphagia scale | baseline/ change from baseline when electrical stimulation applied(the object of this study is to know the temporary change of dysphagia when stimulating with 4ch NMES.
  total score 100 from 0, 100 is worst outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ju Seok Ryu, M.D. PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Kyungji-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim J, Lee JC, Jang EG, Choi SY, Seo KH, Lee SY, Park D, Oh BM, Seo HG, Ryu JS. Kinematic mechanism of the rehabilitative effect of 4-channel NMES: post-hoc analysis of a prospective randomized controlled study. Sci Rep. 2023 Aug 18;13(1):13445. doi: 10.1038/s41598-023-40359-3. PMID 37596323
- [Derived] Seo KH, Jang J, Jang EG, Park Y, Lee SY, Kim BR, Park D, Park S, Hwang H, Kim NH, Oh BM, Seo HG, Lee JC, Ryu JS. Clinical effectiveness of the sequential 4-channel NMES compared with that of the conventional 2-channel NMES for the treatment of dysphagia in a prospective double-blind randomized controlled study. J Neuroeng Rehabil. 2021 May 31;18(1):90. doi: 10.1186/s12984-021-00884-6. PMID 34059092